CLINICAL TRIAL: NCT04559399
Title: Smiley Face Shaped Rod Technique Versus Instrumented Posteriolateral Fusion in Treatment of Isthmic Lumbar Spondylolisthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Najib Mohammed AL-shaea, Principal Investigator,assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: isthmic spondylolisthesis
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Isthmic Spondylolisthesis

STUDY DESIGN:
Intervention Model Description: all patients confirmed diagnosis and including criteria of intervention divided randomly in to 2 groups,control group include patients treat by transpedical screw and rod fixation and experimental group include patients treats smiley face rod technique and then clinical and radiological follow up for 6 month.
  the varibals that will be measure are:
  1. intraoperative variables :length of wound,blood loss and time of operation.
  2. clinical outcome:pain and disability
  3. radiological variables :fusion and degenerative of the adjacent level
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: smiley face shape rod — For treatment of isthmic spondylolithesis a transpedical screws for the same level and rod revolve around spinal process to stabilization of pars interarticularis of the same segment after removes bone at the margine of defects pars till reach to healthy bleed margine then put bone graft at the defect then stablizing pars and bone graft by rods.

SUMMARY:
Aim of research is to investigates clinical, surgical and radiological outcome of vertebral pars intetarticularis repair by used smile face shape rod technique and bone grafting and comparing that with posteriolateral fusion with used traditional transpedical screw and rod fixation in management of isthmic spondylistheisis

DETAILED DESCRIPTION:
Isthmic spondylolisthesis is considered to represent a fatigue fracture of the pars interarticularis of the neural arch, The clinical symptom is activity-related back pain in young and athletic patients . The cause of Isthmic spondylolisthesis in these patients is repetitive stress of the pars interarticularis with subsequent microfracture, which in turn may lead to a bony defect and cause progressive spondylolisthesis in up to 25% of cases. Surgical intervention is indicated for patients who are not responsive despite adequate period of conservative management such as activity modification , physical therapy, and occasionally bracing .

Techniques for repair of a pars defect include Scott wiring , a Buck screw , a pedicle screw and hook , multiple segment fixations or a U-rod . After repair, radiographic healing rates range from 67 percent to 90 percent; asymptomatic and return to sports rates range from 80 percent to 90 percent.

These methods have achieved variable success .In Buck screw fusion surgery,it is not effect on flexion and axial rotation of the spine but bone healing is compromised.

Stabilization with wiring and titanium cable had less success rate than other methods and requires the use of lumbar brace or prolonged immobilization.

The pedicle screw-vertebral plate hook system may complicated by injury to the dural sac or nerves ensues.

Multiple segment fixation with pedicle screws and rods has good success of stabilization but it is effect on flexion and axial rotation of the spine, and may cause degenerative change in adjacent normal segments.

Smiley face shaped rod technique is new method used for repair of isthmic spodylolisthesis using pedical screw on effected segment and smiley face rod revolve around spinal process to stabilization of pars interarticularis of the same segment so it preserve axial rotation and flexion of spin also avoid degenerative change in adjacent levels.

ELIGIBILITY:
Inclusion Criteria:

1. age above 18 years old
2. Both sex
3. failure of conservative treatment for 3months
4. fit for surgery

Exclusion Criteria:

1. age less than 18
2. Not fit for surgery
3. pathological fracture of pars
4. assosciated pathology like disc degeneration, spinal canal stenosis, spondylolisthesis grad 2,3and 4

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
change pain | pain assess one week postoperation
  assessment of pain change one week postoperation by using visual analog scale (AVS) and MacNabs chart to assess degree of change
radiological fusion of pars defect | 6 month postoperative
  using CT scan for fusion percentage assess at 6 month of postoperation.

REFERENCES:
- [Background] Standaert CJ, Herring SA. Spondylolysis: a critical review. Br J Sports Med. 2000 Dec;34(6):415-22. doi: 10.1136/bjsm.34.6.415. PMID 11131228
- [Background] Widi GA, Williams SK, Levi AD. Minimally invasive direct repair of bilateral lumbar spine pars defects in athletes. Case Rep Med. 2013;2013:659078. doi: 10.1155/2013/659078. Epub 2013 Apr 30. PMID 23737800
- [Background] Debnath UK, Freeman BJ, Gregory P, de la Harpe D, Kerslake RW, Webb JK. Clinical outcome and return to sport after the surgical treatment of spondylolysis in young athletes. J Bone Joint Surg Br. 2003 Mar;85(2):244-9. doi: 10.1302/0301-620x.85b2.13074. PMID 12678361
- [Background] Bell DF, Ehrlich MG, Zaleske DJ. Brace treatment for symptomatic spondylolisthesis. Clin Orthop Relat Res. 1988 Nov;(236):192-8. PMID 3180570
- [Background] Bonnici AV, Koka SR, Richards DJ. Results of Buck screw fusion in grade I spondylolisthesis. J R Soc Med. 1991 May;84(5):270-3. doi: 10.1177/014107689108400509. PMID 2041003
- [Background] Herman MJ, Pizzutillo PD, Cavalier R. Spondylolysis and spondylolisthesis in the child and adolescent athlete. Orthop Clin North Am. 2003 Jul;34(3):461-7, vii. doi: 10.1016/s0030-5898(03)00034-8. PMID 12974495
- [Background] Karatas AF, Dede O, Atanda AA, Holmes L Jr, Rogers K, Gabos P, Shah SA. Comparison of Direct Pars Repair Techniques of Spondylolysis in Pediatric and Adolescent Patients: Pars Compression Screw Versus Pedicle Screw-Rod-Hook. Clin Spine Surg. 2016 Aug;29(7):272-80. doi: 10.1097/BSD.0b013e318277cb7d. PMID 23075858
- [Background] Chen XS, Zhou SY, Jia LS, Gu XM, Fang L, Zhu W. A universal pedicle screw and V-rod system for lumbar isthmic spondylolysis: a retrospective analysis of 21 cases. PLoS One. 2013 May 17;8(5):e63713. doi: 10.1371/journal.pone.0063713. Print 2013. PMID 23691090